CLINICAL TRIAL: NCT02101450
Title: Evaluation of the Effects of Extra-abdominal Removal of the Placenta During Cesarean Section on the Amount of Bleeding Into the Abdominal Cavity.
Brief Title: Extra-abdominal Removal of Placenta During CS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Baris KAYA, OBSTETRICS AND GYNECOLOGY CONSULTANT, MD, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KAYA-2013-1
Record Dates: First submitted 2014-03-15; First posted 2014-04-02 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: the Influence of Intra- vs Extra-abdominal Removal of Placenta; Duration of Operation; the Amount of Aspirated Fluid During the Operation; Difference Between Pre- and Post-operative CBC
Keywords: extra-abdominal; intra-abdominal; removal of placenta; cesarean section; bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intra-abdominal removal of the placenta (No Intervention): The uterus will be left in the abdominal cavity and the placenta will be manually removed with uterine massage as soon as possible. After removal of the placenta, the uterus will be dragged out of the abdominal cavity. The cesarean incision will be sutured with no. 1 Vicryl ®. Uterus will be replaced in the abdominal cavity. Intra-abdominal cavity will be cleaned by aspirator and mounted-gauze tampon. The weight of the placenta will be measured. The weight of the gauze tampons will be measured with gravimetric method before and after use.
- Extra-abdominal removal of the placenta (Experimental): No drug or device is used. The uterus will be dragged out of the abdominal cavity, prior to removal of the placenta.
  The placenta will be manually removed with uterine massage as soon as possible. The cesarean section will be completed as described in "No intervention" group.
  Interventions: Procedure: Extra-abdominal removal of the placenta

INTERVENTIONS:
Procedure: Extra-abdominal removal of the placenta — The uterus will be dragged out of the abdominal cavity, prior to removal of the placenta.
  Arms: Extra-abdominal removal of the placenta
Procedure: Extra-abdominal removal of the placenta — The placenta will be manually removed extra-abdominally, with uterine massage as soon as possible.
  Arms: Extra-abdominal removal of the placenta
Procedure: Extra-abdominal removal of the placenta — The cesarean incision will be sutured with no. 1 Vicryl ®.
  Arms: Extra-abdominal removal of the placenta
Procedure: Extra-abdominal removal of the placenta — Uterus will be replaced in the abdominal cavity.
  Arms: Extra-abdominal removal of the placenta

SUMMARY:
During cesarean section, it is important to provide hemostasis as well as to decrease the amount of hemorrhagic fluid and fibrin in the abdominal cavity. Hemorrhagic fluid and fibrin together may cause adhesion formation and therefore postoperative ileus, retardation in regaining the gastrointestinal functions as well as prolongation of the operation itself. Dragging the uterus out of the abdominal cavity during cesarean section before removing the placenta (extra-abdominal removal of the placenta) may decrease the amount of blood flowing into the abdominal cavity during removal of placenta. In this study the investigators aimed to evaluate the influence of intra abdominal vs extra abdominal removal of placenta on duration of operation, the amount of aspirated fluid during the operation, difference between postoperative hemoglobin and hematocrit levels, postoperative pain score, additional need of analgesia, postoperative bowel movements, postoperative endometritis and wound infection.

DETAILED DESCRIPTION:
In this study the investigators will recruit 200 pregnant women; 100 women in the study group and 100 women in the control group. The women will be randomly allocated in two groups. The odd numbered women will be in the study group and even numbered women will be in the control group.

The investigators will perform cesarean section according to the obstetrical indications. Lower segment uterine incision will be used during the cesarean section. After the delivery of the fetus two distinct procedures will be used in the control and study groups.

In the control group, the uterus will be left in the abdominal cavity and the placenta will be manually removed with uterine massage as soon as possible. After removal of the placenta, the uterus will be dragged out of the abdominal cavity. The cesarean incision will be sutured with no. 1 Vicryl ®. Uterus will be replaced in the abdominal cavity. Intra-abdominal cavity will be cleaned by aspirator and mounted-gauze tampon. The weight of the placenta will be measured. The weight of the gauze tampons will be measured with gravimetric method before and after use.

In the study group, at first, the uterus will be dragged out of the abdominal cavity, prior to removal of the placenta. The placenta will be manually removed with uterine massage as soon as possible. The cesarean incision will be sutured with no. 1 Vicryl ®. Uterus will be replaced in the abdominal cavity. Intra-abdominal cavity will be cleaned by aspirator and mounted-gauze tampon. The weight of the placenta will be measured. The weight of the gauze tampons will be measured with gravimetric method before and after use.

In both groups, the abdominal cavity will be closed as appropriate. The vital signs (blood pressure and heart rate) will be monitored. Postoperative blood samples for complete blood count (CBC) will be taken 24 hours after the operation. Bowel movements will be assessed every 6 hours by a stethoscope. Time of the first flatulence will be recorded. Visual Analog Scoring (VAS) survey validated in Turkey will be performed in the postoperative 1. and 2. days. The type and amount of postoperative analgesics will be recorded. The body temperature will regularly be assessed in the first 24. and 48. hours. The presence of fever will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing cesarean section according to the obstetrical indications.

Exclusion Criteria:

* Uterine anomalies such as didelphys, bicornis, etc.
* Placental adhesion anomalies
* Postpartum uterine hemorrhage (>500 ml)
* Polyhydramnios
* Uterine atony
* Women with known coagulation disorders
* Abnormal preoperative APTT, PT and INR

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The amount of aspirated fluid during the cesarean section | 3 months
  The amount of aspirated fluid during the cesarean section in mililiters

SECONDARY OUTCOMES:
Difference between preoperative and postoperative hemoglobin levels | 3 months
  Difference between preoperative and postoperative hemoglobin levels expressed as g/dL
The weight of the gauze before and after use in cesarean section | 3 months
  The weight of the gauze before and after use in cesarean section, described in miligrams

CONTACTS AND LOCATIONS:
Overall Officials: Baris Kaya, MD, Principal Investigator — Near East University, Obstetrics and Gynecology, Lefkosa-TRNC, Mersin 10, Turkey
Locations (1):
- Near East University, Obstetrics and Gynecology, Mersin, Trnc, Turkey (Türkiye)